CLINICAL TRIAL: NCT03841552
Title: Efficacy of Augmented Feedback on Lumbar Postural and Movement Control During Physiotherapy and Home Exercise - A Randomized Controlled Pilot Trial
Brief Title: Efficacy of Augmented Feedback on Lumbar Postural and Movement Control During Physiotherapy and Home Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zurich University of Applied Sciences (Other)
Collaborators: Danube University Krems (Other); MedBase Brunngasse Winterthur (Unknown)
Responsible Party: Principal Investigator, Markus J. Ernst, research associate, Zurich University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KEK-ZH-Nr. 2011-0522
Record Dates: First submitted 2019-02-05; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Low Back Pain
Keywords: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized controlled pilot trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators who collected the outcome data, as well as the statistician were blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Augmented Feedback (Experimental): The exercises were conducted with the aim of improving postural- and movement control and awareness of the lumbar spine in both treatment groups. Both groups received nine 30-minute therapy sessions, during which they performed a series of exercises from an exercise catalogue. The exercises were selected based on their compatibility with the AF-system. Each patient performed impairment-specific exercises. The AF group received additional AF feedback during both the therapy sessions and the home exercise program, by combining the exercises with games designed to target movement control, body awareness, and stabilisation exercises.
  Interventions: Device: Augmented Feedback
- Control Group (Active Comparator): The control group performed the impairment-specific exercises without AF. The control group was able to receive conventional visual feedback, such as use of mirrors, as deemed appropriate by the therapists but no AF.
  Interventions: Other: Control Group

INTERVENTIONS:
Device: Augmented Feedback — An inertial measurement unit (IMU) system is the basis of the augmented feedback (AF) system, where the IMU-system communicates with a laptop using a bluetooth dongle. The corresponding software includes therapeutic games. Movements of the lower back and pelvis by the patient are used to control an avatars movement or the graphical interface in computer exercises. The AF-system provides real-time feedback regarding the patient's performance and helps to rectify incorrect execution of the exercises. The intervention took place at a physiotherapy clinic and in an home environment. In the physiotherapy clinic the patients exercised under the supervision of the physiotherapists. They continued the exercises at home as home exercises.
  Arms: Augmented Feedback
Other: Control Group — Conventional impairment-specific physiotherapy exercises for low back pain patients.The control intervention took place at a physiotherapy clinic and in an home environment. In the physiotherapy clinic the patients exercised under the supervision of the physiotherapists. They continued the exercises at home as home exercises.
  Arms: Control Group

SUMMARY:
Exercise therapy is effective in improving pain experience and disability in patients with non-specific low back pain (NSLBP) and movement/postural control impairments. However, patients often find traditional exercises monotonous and discontinue their execution. Augmented feedback tools (AF) might improve patient adherence and therapy outcomes, but evidence is currently lacking on their effects on movement/postural control. In a pilot randomised controlled trial (RCT) on a population of patients with NSLBP and movement control impairment, treatment with physiotherapy and home exercise supported by AF is compared to traditional physiotherapy and home exercise treatment without AF (control group). The primary outcomes are defined as lumbar movement control and postural control, measured using an inertial measurement system.

ELIGIBILITY:
Inclusion Criteria:

* non specific low back pain for at least four weeks
* at least moderate disability (as indicated by an Oswestry disability index (ODI) > 8% (Mannion et al., 2006))
* low levels of biopsychosocial risk factors (STarT Back Screening tool > 4 points) (Hill et al., 2011)
* at least two positive movement control impairment tests (Luomajoki et al., 2008, Sahrmann, 2002)

Exclusion Criteria:

* specific low back pain
* pain in other areas of the body (e.g. neck, head, thoracic spine or arms)
* vertigo or equilibrium disturbances
* systemic diseases (e.g. tumours and diabetes)
* injuries
* surgeries of the legs within the last six months
* medication affecting postural control
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2013-04-30 (Actual); Study Completion 2013-04-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline ratio of the range of motion (ROM) of the stabilized lumbar spine (ROMLS) over the moving body segment, the hip (ROMHip) | From Baseline to the completion of nine physiotherapy sessions, which are completed after a maximum of five weeks (Swiss standard prescription)
  Movement control was quantified using the ratio of the range of motion (ROM) of the stabilized lumbar spine (ROMLS) over the moving body segment, the hip (ROMHip) during the movement control test (lumbar spine (LS) over the hip)
Changes from Baseline of the mean absolute deviation of lumbar agular displacement | From Baseline to the completion of nine physiotherapy sessions, which are completed after a maximum of five weeks (Swiss standard prescription)
  Postural control was quantified using the mean absolute deviation of lumbar angular displacement (MAD)

CONTACTS AND LOCATIONS:
Locations (1):
- Zurich University of Applied Sciences, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hugli AS, Ernst MJ, Kool J, Rast FM, Rausch-Osthoff AK, Mannig A, Oetiker S, Bauer CM. Adherence to home exercises in non-specific low back pain. A randomised controlled pilot trial. J Bodyw Mov Ther. 2015 Jan;19(1):177-85. doi: 10.1016/j.jbmt.2014.11.017. Epub 2014 Nov 27. PMID 25603757